CLINICAL TRIAL: NCT00335972
Title: Phase 4: The Effects of Dexmedetomidine and Remifentanil on Postoperative Hemodynamics and Pain/Opioids in Patients Undergoing Carotid Endarterectomy
Brief Title: The Effects of Dexmedetomidine and Remifentanil on Carotid Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Closed due to lack of enrollment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 10-27-05
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Carotid Artery Stenosis
Keywords: Carotid Endarterectomy patients
MeSH Terms: conditions — Carotid Stenosis | interventions — Remifentanil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remifentanil (Active Comparator): Remifentanil will be infused throughout surgery at a rate of 0.1-0.2 µg/kg/min. Propofol will be titrated to maintain a BIS value as close to 45 as clinically practical
  Interventions: Drug: Remifentanil
- Dexmedetomidine (Active Comparator): Dexmedetomidine, 0.5-1 µg/kg, will be infused over 20 minutes, immediately followed by an infusion at a rate of 0.2 µg/kg/hr until the end of surgery (For patients in renal failure, the loading dose will be 0.2 µg/kg). The infusion rate will be reduced as necessary to maintain acceptable blood pressure and heart rate. Propofol will be titrated to maintain BIS as close to 45 as clinically practical.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remifentanil — Remifentanil will be infused throughout surgery at a rate of 0.1-0.2 µg/kg/min. Propofol will be titrated to maintain a BIS value as close to 45 as clinically practical
  Arms: Remifentanil
Drug: Dexmedetomidine — Dexmedetomidine, 0.5-1 µg/kg, will be infused over 20 minutes, immediately followed by an infusion at a rate of 0.2 µg/kg/hr until the end of surgery (For patients in renal failure, the loading dose will be 0.2 µg/kg). The infusion rate will be reduced as necessary to maintain acceptable blood pressure and heart rate. Propofol will be titrated to maintain BIS as close to 45 as clinically practical.
  Arms: Dexmedetomidine

SUMMARY:
We propose to test whether intraoperative administration of dexmedetomidine will reduce hemodynamic control in the intra- and post-operative periods and reduces PACU analgesic requirements in patients undergoing carotid endarterectomy.

DETAILED DESCRIPTION:
Remifentanil is an amidopiperidine derivative with unique pharmacokinetic properties. Its steady-state volume of distribution is 30 L (3). Its context-sensitive half life is consistently short (3.2 min), even after prolonged infusion(4). The pharmacokinetic profile of remifentanil is independent of the hepatic (5) and renal function (6). And finally, the recovery profile of remifentanil is excellent with a speedy anesthetic emergence time which is important for a quick and proper neurologic assessment in the early postoperative period.

Remifentanil produces good intraoperative hemodynamic control during intense noxious stimulation like laryngoscopy, endotracheal intubation, and during pinning of the head (8). However, side effects of remifentanil include hypotension and bradycardia (15) intraoperatively, along with apnea(16,17) and hyperalgesia(18) postoperatively which is caused by increasing sensitivity to noxious stimuli. Investigations demonstrate different mechanisms of opioid-induced post-infusion anti-analgesia and secondary hyperalgesia (9). Overall remifentanil is a versatile opioid that is being increasingly used in the operating room.

DEXMEDETOMIDINE (DEX), an alpha-2 adrenoreceptor agonist, is gaining popularity in neuroanesthesia. It has a desirable neurophysiologic profile including neuroprotective characteristics through its effect on α2A receptor subtypes (10). Its hypnotic effect is mediated through the α2 receptors in the locus ceruleus and its analgesic properties are mediated through an effect on the dorsal horn of the spinal cord (11,12). Since it has sympatholytic and antinociceptive properties, it may improve hemodynamic stability at critical moments of neurosurgical stimulation. Dexmedetomidine reduces anesthetic drug and opioid requirements in the perioperative period (13,14). In addition, dexmedetomidine does not affect evoked potential monitoring, (19) making it a favorable anesthetic adjunct in cases in which neurophysiologic monitoring is being used. In recent years, dexmedetomidine has emerged as an effective drug useful in a wide range of anesthesia related areas.

Study Questions We postulate that dexmedetomidine provides better hemodynamic control in the intra- and post-operative periods and reduces PACU analgesic requirements.

Primary Hypothesis 1: Intraoperative dexmedetomidine provides better postoperative analgesia than remifentanil, thus reducing PACU opioid requirements.

Primary Hypothesis 2: Dexmedetomidine causes fewer hemodynamic perturbations than remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult patients (age >50 years) undergoing carotid endarterectomy with general anesthesia.

Exclusion Criteria:

* Receiving another alpha 2-adrenoreceptor agonist;
* Contraindication to dexmedetomidine, including allergy;
* Current hepatic disease (liver function tests > twice upper limit of normal);
* Renal insufficiency, as defined by a creatinine > 2.0 mg/dL;
* Mentally impairment, including dementia or delirium;
* Heart block ;
* Sick sinus syndrome;
* Atrial fibrillation with a low ventricular response (< 50 bpm);
* Absolute or relative hypovolemia;
* Prior stroke;
* Severe left-ventricular dysfunction

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Farag, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remifentanil | Dexmedetomidine
Started | 71 | 71
Completed | 71 | 68
Not Completed | 0 | 3
Not completed — not given treatments | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil | Dexmedetomidine | Total
Number analyzed (Participants) | 71 | 68 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (14) | 56 (14) | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 70
  Male | 34 | 35 | 69
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race-white | 65 | 57 | 122
  Race-other | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Pressure
Time Frame: mean arterial pressure at 15, 30, 45, 60, and 90 minutes after extubation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
mmHg
  at 15 minutes after extubation | 99 (12) | 86 (13)
  at 30 minutes after extubation | 98 (12) | 87 (13)
  at 45 minutes after extubation | 98 (13) | 86 (13)
  at 60 minutes after extubation | 96 (12) | 89 (15)
  at 90 minutes after extubation | 94 (12) | 88 (13)
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Test type: Non-Inferiority or Equivalence — Sample size was based on being able to detect noninferiority on both analgesia (pain score and opioids) and hemodynamic responses, and superiority on at least one of them with 90% power and significance level of 0.025 for each of noninferiority and superiority. For MAP with a noninferiority delta of 7.5 mmHg and expected the SD of 12, we needed a maximum of N= 65 per group. Incorporating the two interim and one final analyses, we thus planned a maximum sample size of N=71/group (N=142 total); p < 0.001, repeated measures ANOVA — Noninferiority confidence intervals are 95% (alpha of 0.05/2=0.025 in direction of interest). Bonferroni correction was used for superiority testing and 97.5% CI were reported; Mean Difference (Net) = -9, 95% CI 2-sided [-13 to -5] — mean difference: Dexmedetomidine arm - Remifentanil arm
Statistical Analysis 2: Comparison: Remifentanil vs Dexmedetomidine; superiority test; Test type: Superiority or Other; p < 0.001, repeated measures ANOVA model — Bonferroni correction was used for superiority testing since superiority on either hemodynamics or pain control would be interpreted as Dex better than Remi (alpha=0.0125 = 0.025/2, 97.5% CI); Mean Difference (Net) = -9, 97.5% CI 2-sided [-13 to -4] — mean difference: dexmedetomidine arm - remifentanil arm

2. Primary Outcome: Visual Analogue Scale (VAS) Pain Score
Description: Using a ruler, the score is determined by measuring the distance on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10. 0 = no pain and 10 = worst
Time Frame: pain score measured at 15, 30, 45, 60, and 90 minutes after extubation
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
cm
  at 15 minutes after extubation | 5.4 (3.4) | 2.6 (3.4)
  at 30 minutes after extubation | 5.3 (2.8) | 2.8 (3.2)
  at 45 minutes after extubation | 5.0 (2.4) | 3.1 (3.0)
  at 60 minutes after extubation | 4.9 (2.6) | 2.9 (2.7)
  at 90 minutes after extubation | 4.8 (2.4) | 2.9 (2.8)
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Test type: Non-Inferiority or Equivalence — Sample size was based on being able to detect noninferiority on both analgesia (pain score and opioids) and hemodynamic responses, and superiority on at least one of them with 90% power and significance level of 0.025 for each of noninferiority and superiority. For VRS pain, the standard deviation (SD) was expected to be about 1.75, such that with a noninferiority delta of 1, we needed a maximum of N= 66 per group; p < 0.001, repeated measures ANOVA model — noninferiority confidence intervals are 95% (alpha of 0.05/2=0.025 in direction of interest); Mean Difference (Net) = -1.9, 95% CI 2-sided [-2.7 to -1.1] — mean difference: Dexmedetomidine arm - Remifentanil arm
Statistical Analysis 2: Comparison: Remifentanil vs Dexmedetomidine; superiority test; Test type: Superiority or Other; p < 0.001, repeated measures ANOVA model — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -1.9, 97.5% CI 2-sided [-2.8 to -0.9] — mean difference: dexmedetomidine arm - remifentanil arm

3. Primary Outcome: Intravenous Morphine Equivalents During Post-anesthesia Care Unit (PACU) After Surgery
Description: intravenous morphine equivalents (mg)
Time Frame: During Post-anesthesia care unit after surgery,an average of 4 hours
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Remifentanil | Dexmedetomidine
Number analyzed (Participants) | 71 | 68
mg | 10 [7 to 15] | 5 [0 to 10]
Statistical Analysis 1: Comparison: Remifentanil vs Dexmedetomidine; Test type: Non-Inferiority or Equivalence — Sample size was based on being able to detect noninferiority on both analgesia (pain score and opioids) and hemodynamic responses, and superiority on at least one of them with 90% power and significance level of 0.025 for each of noninferiority and superiority.we needed a maximum of N= 65 per group. We assumed for opioids that the coefficient of variation (SD/mean) was about 0.4, resulting in a similar sample size (64/group) with noninferiority deltas of 20% of the observed mean; p < 0.001, Wilcoxon (Mann-Whitney) — noninferiority confidence intervals are 95% (alpha of 0.05/2=0.025 in direction of interest); Mean Difference (Net) = -5, 95% CI 2-sided [-10 to -5] — mean difference: Dexmedetomidine arm - Remifentanil
Statistical Analysis 2: Comparison: Remifentanil vs Dexmedetomidine; superiority; Test type: Superiority or Other; p < 0.001, repeated measures ANOVA model — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -5, 97.5% CI 2-sided [-10 to -3] — mean difference: dexmedetomidine arm - remifentanil arm

ADVERSE EVENTS:
Time Frame: during Post-anesthesia care unit after surgery
Arm/Group | Remifentanil | Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/68
Other Adverse Events (participants affected / at risk) | 0/71 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No